CLINICAL TRIAL: NCT00906035
Title: The Vascular Biology of Dipyridamole in Peripheral Arterial Disease (PAD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not enroll subjects who met the stringent inclusion/exclusion criteria.
Sponsor: University of Pennsylvania (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 706469; 0821
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; PAD; Claudication; Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Peripheral Vascular Diseases | interventions — Dipyridamole; Aspirin; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dipyridamole 200mg and Aspirin 25mg bid (Active Comparator): All subjects in this arm will take their assigned medication for 180 days and complete study visits on Day 1(Baseline), 30, 90 and 180. All subjects will bring a 24 hour urine collection and arrive in a fasting state on all visit days for a blood draw after which they will receive breakfast. After assessing vitals, Adverse Event status and medication compliance, they will be escorted to the vascular labs for Doppler Ultrasound and Near Infrared Spectroscopy. (NIRS) of the legs.
  Interventions: Drug: Dipyridamole 200mg and Aspirin 25mg bid:
- Dipyridamole 200 mg bid (Active Comparator): All subjects in this arm will take their assigned medication for 180 days and complete study visits on Day 1(Baseline), 30, 90 and 180. All subjects will bring a 24 hour urine collection and arrive in a fasting state on all visit days for a blood draw after which they will receive breakfast. After assessing vitals, Adverse Event status and medication compliance, they will be escorted to the vascular labs for Doppler Ultrasound and Near Infrared Spectroscopy. (NIRS) of the legs.
  Interventions: Drug: Dipyridamole 200 mg bid
- Aspirin 25 mg bid (Active Comparator): All subjects in this arm will take their assigned medication for 180 days and complete study visits on Day 1(Baseline), 30, 90 and 180. All subjects will bring a 24 hour urine collection and arrive in a fasting state on all visit days for a blood draw after which they will receive breakfast. After assessing vitals, Adverse Event status and medication compliance, they will be escorted to the vascular labs for Doppler Ultrasound and Near Infrared Spectroscopy (NIRS) of the legs.
  Interventions: Drug: Aspirin 25 mg bid

INTERVENTIONS:
Drug: Dipyridamole 200mg and Aspirin 25mg bid: — All subjects will receive their randomly assigned study medication to be taken each morning and evening approximately 8am and 8 pm for the 180 day duration of the study.
  Other Names: Persantine
  Arms: Dipyridamole 200mg and Aspirin 25mg bid
Drug: Dipyridamole 200 mg bid — All subjects will receive their randomly assigned study medication to be taken each morning and evening approximately 8am and 8 pm for the 180 day duration of the study.
  Other Names: Persantine
  Arms: Dipyridamole 200 mg bid
Drug: Aspirin 25 mg bid — All subjects will receive their randomly assigned study medication to be taken each morning and evening approximately 8am and 8 pm for the 180 day duration of the study.
  Arms: Aspirin 25 mg bid

SUMMARY:
This research study will evaluate the effects of aspirin and dipyridamole alone and in combination on the blood flow in the vessels of the legs. We will examine how these medications are able to inhibit the clotting of platelets in the vessels of patients with PAD, and thereby affect the blood flow in the legs. Platelets are cells in the blood that have the ability to adhere to each other to form clots.

DETAILED DESCRIPTION:
Dipyridamole has been reformulated to guarantee systemic bioavailability and steady state levels compatible with inhibition of platelet aggregation ex vivo (1). This newly formulated dipyridamole has been shown to roughly equal in efficacy to low dose aspirin in the secondary prevention of stroke and the drug combination seems roughly additive (2). The present study is designed to explore two potential mechanisms which have been linked to dipyridamole action on the vessel wall; modulation of vascular eicosanoid generation and prevention of oxidant stress (3). We shall address the hypothesis that dipyridamole affects these systems in patients with PAD. These individuals have disordered platelet-vascular interactions, as reflected by increased generation of thromboxane, an index of platelet activation and of prostacyclin, probably a homeostatic response to traumatic and chemical stimulation of the endothelium (4,5). Furthermore, we shall assess the functional consequences of dipyridamole action, alone and in combination with aspirin compared with aspirin alone on local measurements of flow and oxygenation, including exercise tolerance, Doppler Ultrasound and Near Infrared Spectroscopy (NIRS). Lipid peroxidation will be quantified based on mass spectrometric analysis of the major urinary isoprostane, 8,12-iso-iPF2a-VI (6,7).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 79
* Women of child bearing potential using a medically acceptable method of birth control (oral/transdermal/vaginal hormonal contraception, depo-provera injection, IUD, condom with spermicide, progestin implant, tubal ligation, oophorectomy, TAH) or abstinence.
* Capacity for giving written consent
* Diagnosis of PAD by:

  * previous angiogram (>0.5 stenosis of a peripheral artery)
  * ankle-brachial index (ABI) of systolic pressure <0.80
  * previous peripheral revascularization
* Smokers who smoke < 10 cigarettes / day

Exclusion Criteria:

* Female subjects who are pregnant or nursing a child.
* Prior bleeding event related to drug therapy
* History of gastrointestinal ulceration
* History of known dipyridamole and/or aspirin allergy or intolerance
* History of coagulation, bleeding or blood disorders.
* Recent history of myocardial infarction or stroke in the previous 6 months
* Resting blood pressure of <110mmHg systolic or <60mmHg diastolic or of >165mmHg systolic or >95mmHg diastolic
* Patients with active infection as documented by abnormal laboratory tests at screen
* Concomitant serious illness, such as cancer, as per the principal investigator's discretion
* Current use of steroids for a chronic disease process
* Presence of ischemic leg ulcers
* History of contact allergies to the metal leads of the NIRS
* History of drug or alcohol abuse within the last 6 months.
* Subject who has received an experimental drug and/or used an experimental device within 30 days of screening.
* Subject who has donated ≥ one pint of blood within 8 weeks prior to screen.
* Use of aspirin for 2 weeks prior to the study
* Use of any other NSAID or COX-inhibitor for one week prior to the start of the study
* Use of any antioxidant vitamin for 2 weeks prior to the start of the study
* Use of plavix, pletal or trental for one week prior to the start of the study
* Use of acetaminophen for one week prior to each study visit
* Use of alcohol, caffeine or high fat foods for 24 hours prior to each study visit
* Has smoked any cigarettes for 24 hours prior to each study visit
* Platelet aggregation blood test less than 60 percent at Visit 1

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-09; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garret A FitzGerald, MD, Principal Investigator — University of Pennsylvania; Emile R Mohler, MD, Principal Investigator — University of Pennsylvania; Tilo Grosser, MD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Presbyterian Hospital, 51 N. 39th St., Philadelphia, Pennsylvania
  - Translational Research Ctr.,3400 Civic Center Blvd, Building 421, 10th floor, Room 421, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dipyridamole 200mg and Aspirin 25mg Bid | Dipyridamole 200 mg Bid | Aspirin 25 mg Bid
Started | 8 | 9 | 8
Completed | 6 (One Drop-Out; SAE day before Visit 1 and One subject Withrew prior to visit 1) | 6 (2 subjects Withdrew after Visit 1 and 1 subject Withdrew shortly after Visit 1due to an AE) | 8
Not Completed | 2 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dipyridamole 200mg and Aspirin 25mg Bid | Dipyridamole 200 mg Bid | Aspirin 25 mg Bid | Total
Number analyzed (Participants) | 8 | 9 | 8 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 3
  >=65 years | 7 | 8 | 7 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 6
  Male | 7 | 7 | 5 | 19
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: The Present Study is Designed to Explore Two Potential Mechanisms Which Have Been Linked to Dipyridamole Action on the Vessel Wall; Modulation of Vascular Eicosanoid Generation and Prevention of Oxidant Stress.
Description: No analysis could be performed due to the insufficent number of participants enrolled. Data were not collected due to study termination related to the difficulty finding participants that matched the inclusion/exclusion criteria.
Time Frame: Predose and dosing days 30, 90 and 180
Population: Data could not collected due to study termination related to the difficulty finding participants that matched the inclusion/exclusion criteria. Data could not be analyzed due to insufficient number of participants enrolled.
Arm/Group | Dipyridamole 200mg and Aspirin 25mg Bid | Dipyridamole 200 mg Bid | Aspirin 25 mg Bid
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Assess the Functional Consequences of Dipyridamole Action, Alone and in Combination With Aspirin Compared With Aspirin Alone on Local Measurements of Flow and Oxygenation. Blood Flow Reporting to Added Table.
Description: Done by doppler ultrasound. Data could not be analyzed due to insufficient number of participants enrolled. Data were not collected due to study termination related to the difficulty finding participants that matched the inclusion/exclusion criteria.
Time Frame: Predose and dosing days 30, 90 and 180.
Population: Data could not be analyzed due to insufficient number of participants enrolled. Data were not collected due to study termination related to the difficulty finding participants that matched the inclusion/exclusion criteria.
Arm/Group | Dipyridamole 200mg and Aspirin 25mg Bid | Dipyridamole 200 mg Bid | Aspirin 25 mg Bid
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Assess the Functional Consequences of Dipyridamole Action, Alone and in Combination With Aspirin Compared With Aspirin Alone on Local Measurements of Flow and Oxygenation. Reporting Blood Oxygenation.
Description: Reporting blood oxygenation. Data could not be analyzed due to insufficient number of participants enrolled. Difficulty finding participants who fit into the inclusion/exclusion criteria.
Time Frame: Predose and dosing days 30, 90 and 180.
Population: as for outcome 2
Arm/Group | Dipyridamole 200mg and Aspirin 25mg Bid | Dipyridamole 200 mg Bid | Aspirin 25 mg Bid
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Dipyridamole 200mg and Aspirin 25mg Bid | Dipyridamole 200 mg Bid | Aspirin 25 mg Bid
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/9 | 1/8
Other Adverse Events (participants affected / at risk) | 5/8 | 4/9 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dipyridamole 200mg and Aspirin 25mg Bid (N=8) | Dipyridamole 200 mg Bid (N=9) | Aspirin 25 mg Bid (N=8)
Cardiac catherization of the pelvis (Cardiac disorders) | 1 (1) | 0 | 0
Chest pain (Cardiac disorders) | 0 | 0 | 1 (3)
Surgical removal of renal tumor (Surgical and medical procedures) | 1 (1) | 0 | 0
balloon angioplasty left leg (Surgical and medical procedures) | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dipyridamole 200mg and Aspirin 25mg Bid (N=8) | Dipyridamole 200 mg Bid (N=9) | Aspirin 25 mg Bid (N=8)
intermittent claudication (Vascular disorders) | 2 | 3 | 2
Angina (Cardiac disorders) | 1 | 0 | 1
Diarrhea (General disorders) | 0 | 1 | 1
Headache (General disorders) | 2 | 0 | 1

LIMITATIONS AND CAVEATS:
Study encountered difficulty while attempting to find subjects who met all inclusion/exclusion criteria."0" indicated because no analysis was done on samples obtained. Data could not be analyzed due to insufficient number of participants enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No